CLINICAL TRIAL: NCT02970396
Title: Self-management for People With Epilepsy and a History of Negative Health Events (SMART)
Brief Title: Self-management for People With Epilepsy and a History of Negative Health Events
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Martha Sajatovic, MD, Professor, Case Western Reserve University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-14-07
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Self-Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMART Intervention (Active Comparator): Participants (a total of 120 individuals) will be randomly assigned to either SMART (N=60) or the wait-list control (N= 60), in a 1:1 ratio.
  Interventions: Behavioral: self-management
- Wait-list (Active Comparator): Participants assigned to the wait-list will start the SMART intervention 6 months following randomization.
  Interventions: Behavioral: self-management

INTERVENTIONS:
Behavioral: self-management

SUMMARY:
This is an investigation of adult individuals with epilepsy, and involves educational and behavioral interventions intended to enhance treatment adherence and self-management.

The investigators are adapting a self-management intervention that they developed in a previous study to individuals with epilepsy and a history of negative health events (NHEs), such as accidents and emergency department (ED) visits, diminished quality of life and poor mental well-being. The intervention "Self-management for people with epilepsy and a history of negative health events (SMART)" is intended to reduce NHEs and improve quality of life in people with epilepsy associated with historically disadvantaged groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy
* Negative health event within the last 6 months
* Able to provide written consent and participate in study procedures

Exclusion Criteria:

* Immediate risk of self-harm
* Dementia
* Pregnancy
* Unable to read/understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-09; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in number of negative health events | baseline, 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States